CLINICAL TRIAL: NCT04046926
Title: Relapse in Anorexia Nervosa: a Prospective Longitudinal Study
Brief Title: Relapse in Anorexia Nervosa. A Cohort Study
Status: Completed | Type: Observational
Sponsor: Villa Garda Hospital (Other)
Responsible Party: Principal Investigator, Riccardo Dalle Grave, Director of the Department of Eating and Weight Disorders, Villa Garda Hospital
Other Study IDs: VillaGH
Record Dates: First submitted 2018-12-06; First posted 2019-08-06 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-09

CONDITIONS: Anorexia Nervosa
Keywords: anorexia nervosa; relapse; inpatient; cognitive behavioral therapy; prospective study
MeSH Terms: conditions — Anorexia Nervosa; Recurrence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The hospitalization in patients with anorexia nervosa has often a short-term success, as weight is restored to a healthy level, but high percentage of patients relapse during the first year following the discharge. Starting from the observation that the relapse rate is lower in outpatient than in inpatient settings, the investigators hypothesized that the reason of this difference is the nature of inpatient treatment and post-inpatient therapy. For this reason, different procedures and strategies have been implemented during hospitalization to reduce the relapse after discharge. The aim of the study was to assess the time and the percentage of relapse after inpatient discharge and at follow-up.

DETAILED DESCRIPTION:
Anorexia nervosa is considered one of the most difficult to treat mental disorders and often treatment outcomes are unsatisfactory. Outpatient treatment is the ideal choice for the treatment of anorexia nervosa, but a large subgroup of patients (50-60%) does not respond to outpatient treatments and need more intensive care, such as hospital rehabilitation. The hospitalization has often a short-term success, as weight is restored to a healthy level, but high percentage of patients relapse during the first year following the discharge. Strategies to limit the post-hospitalization relapse rate are now focused on assessing the effectiveness of different treatments given after discharge. Our group, after evaluating the results of a controlled study, used another strategy. Starting from the observation that the relapse rate is lower in outpatient than in inpatient settings, the investigators hypothesized that the reason of this difference is the nature of inpatient treatment and post-inpatient therapy. For this reason, different procedures and strategies have been implemented during hospitalization to reduce the relapse after discharge.

The primary outcome of interest is the proportion of patients who relapse after discharge from hospitalization. For the calculation of the sample size a 95% confidence interval was established, an expected prevalence of 40% and a desired accuracy of 10%. Based on these premises, it is necessary to have a group of "completers" at 60 weeks of follow-up of 92 patients. To calculate the initial sample needed to generate 92 patients at 60 weeks of follow-up, the investigators considered the attrition rate during treatment (set at 13%) and a subsequent attrition rate at follow-ups (set at 10%). This calculation produces a result of an initial sample of 118 patients.

The frequency and time of relapse will be evaluated using Kaplan-Meier survival analysis. Cox proportional hazards regression analysis will be used to examine the role of predictive variables in predicting time to relapse. Univariate Cox regressions and multivariate Cox regressions will be used to evaluate the potentially predictive variables at baseline, during the treatment process, at the end of therapy and during post-discharge.

ELIGIBILITY:
Inclusion Criteria:

1. Female
2. Age >= 13 years and <= 65 years
3. Meeting diagnostic criteria for anorexia nervosa at inpatient admission
4. Full response (i.e., Body Mass Index (BMI) >= 18.5 kg/m2 and Eating Disorder Examination Questionnaire (EDE-Q) global score < 2.77) at discharge
5. Written informed consent

Exclusion Criteria:

1. Acute psychotic disorders
2. Active substance abuse
3. Meeting diagnostic criteria for bulimia nervosa
4. Medical complication that may hamper the interpretation of results (medical condition that causes weight changes)
5. Absence of medical treatment (drugs) that may hamper the interpretation of results
6. Pregnancy or plan to get pregnant

Ages: 13 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The sample includes patients with anorexia nervosa who will be recruited from consecutive referrals to the eating disorder inpatient unit of Villa Garda Hospital (Northern Italy).
Sampling Method: Probability Sample
Enrollment: 118 (Actual)
Dates: Start 2020-05-01 (Actual); Primary Completion 2024-07-01 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Good BMI outcome | 40 weeks after inpatient admission (corresponding to 20 weeks after discharge)
  Body Mass Index >= 18.5 kg/m2

SECONDARY OUTCOMES:
Relapse | 40 weeks after inpatient admission (corresponding to 20 weeks after discharge)
  To evaluate the relapse, investigators need to consider patients with full response at discharge of inpatient treatment (i.e. after 20 weeks from admission) that relapse during the following 20 weeks (i.e 40 weeks after inpatient admission).
  So, the criteria for the relapse are:
  * full response after 20 weeks of inpatient treatment AND
  * underweight BMI (i.e. BMI < 18.5 kg/m2) AND/OR
  * high level of eating disorder psychopathology (i.e. EDE-Q ≥ 2.77)
Full Response | 40 weeks after inpatient admission (corresponding to 20 weeks after discharge)
  To evaluate the full response in underweight eating disorder patients the investigators need to evaluate both the reaching a non-underweight BMI and an eating disorder psychopathology similar to non-clinical cases.
  To evaluate the eating disorder psychopathology the investigators used the Eating Disorder Examination Questionnaire (EDE-Q). The EDE-Q global score range from 0 to 6.
  The criteria for the Full Response are the following:
  * Body Mass Index >= 18.5 kg/m2 AND
  * Eating Disorder Examination Questionnaire (EDE-Q) global score < 2.77.

CONTACTS AND LOCATIONS:
Overall Officials: Riccardo Dalle Grave, MD, Principal Investigator — Department of Eating and Weight Disorders, Villa Garda Hospital
Locations (1):
- Department of Eating and Weight Disorders, Villa Garda Hospital, Garda, Italy, Italy

REFERENCES:
- [Background] Berends T, Boonstra N, van Elburg A. Relapse in anorexia nervosa: a systematic review and meta-analysis. Curr Opin Psychiatry. 2018 Nov;31(6):445-455. doi: 10.1097/YCO.0000000000000453. PMID 30113325
- [Background] Bardone-Cone AM, Harney MB, Maldonado CR, Lawson MA, Robinson DP, Smith R, Tosh A. Defining recovery from an eating disorder: Conceptualization, validation, and examination of psychosocial functioning and psychiatric comorbidity. Behav Res Ther. 2010 Mar;48(3):194-202. doi: 10.1016/j.brat.2009.11.001. Epub 2009 Nov 13. PMID 19945094